CLINICAL TRIAL: NCT02580513
Title: Impact of Circadian Misalignment on Insulin Sensitivity
Brief Title: Circadian Misalignment and Insulin Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: NL54897.068.15
Record Dates: First submitted 2015-10-14; First posted 2015-10-20 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Diabetes Mellitus, Type 2; Insulin Resistance
Keywords: Circadian Rhythm; Circadian Misalignment; Insulin Sensitivity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): 3 days with normal circadian alignment.
- Circadian Misalignment (Experimental): 3.5 days in which the subjects will undergo a maximal circadian misalignment of 12 hours by means of a midday nap during the second day, and a subsequent start of a new normal wake period, shifted 12 hours.
  Interventions: Behavioral: Circadian Misalignment

INTERVENTIONS:
Behavioral: Circadian Misalignment
  Arms: Circadian Misalignment

SUMMARY:
This study will evaluate the effect of circadian misalignment on insulin sensitivity in healthy lean subjects in a randomized cross-over design. Subjects will be admitted to the research facility for two study periods of 3 and 3.5 days. In one of the study periods, the behavioral cycle will be shifted by 12 hours. Insulin sensitivity will be measured with a hyperinsulinemic euglycemic clamp.

DETAILED DESCRIPTION:
Recent evidence shows that misalignment of the circadian rhythm (e.g. by rotating shift work) impairs glucose metabolism markedly, possibly by decreasing insulin sensitivity in peripheral tissues and liver. Nowadays our society is indispensably connected to a lifestyle that allows wakefulness at every time of the 24 hours cycle. Social jetlag is a phenomenon that affects a large part of the general population, thus circadian misalignment extends far beyond those who are on a shift work schedule. Therefore, decreased insulin sensitivity in individuals affected by circadian misalignment may help to explain the increased prevalence of T2DM in night shift workers that has been found in epidemiological studies.

The study is an interventional randomized crossover trial in which each subject serves as it owns control. For the study, the investigators ask the subjects to participate in two study periods, one of 3 days length (control condition) and the other of 3.5 days length (misalignment condition). During the 3.5 day misalignment condition, subjects will shift their day-night rhythm by 12 hours, which will lead to maximal circadian misalignment. Insulin sensitivity will be measured by a hyperinsulinemic euglycemic clamp. Secondary parameters will include ex-vivo skeletal muscle mitochondrial function and whole-body energy metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian
* Healthy (as determined by dependent physician based on medical questionnaire)
* Male
* Age: 18-35 years
* Normal BMI (18-25 kg/m2)
* Regular sleeping time (normally 7 - 9h daily)
* Habitual bedtime at 11 PM ± 2 hours

Exclusion Criteria:

* Extreme early bird or extreme night person
* Heavily varying sleep-wake rhythm
* Shiftwork during last 3 months
* Travel across >1 time zone in the last 3 months
* Engagement in exercise > 3 hours total per week
* Using > 400mg caffeine daily
* Smoking
* Unstable body weight (weight gain or loss > 3kg in the last 3 months)
* Significant food allergies/intolerance (seriously hampering study meals)
* Participation in another biomedical study within 1 month before the first study visit
* Claustrophobia
* Medication use hampering the study (as determined by responsible physician)
* Recent blood donation.
* Any contra-indication to the telemetric pill:
* Any acute condition, exacerbation of chronic condition, or medical history that would in the investigator's opinion interfere with the study

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2016-01; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Insulin Sensitivity | 2 days after circadian misalignment and matched time in control arm.
  Measured with hyperinsulinemic euglycemic clamp

SECONDARY OUTCOMES:
Oxidative glucose disposal | 2 days after circadian misalignment and matched time in control arm.
Non-oxidative glucose disposal | 2 days after circadian misalignment and matched time in control arm.
Skeletal muscle mitochondrial function | 1 and 2 days after circadian misalignment and matched times in control arm
  Measured with high-resolution respirometry on permeabilized muscle fibers after muscle biopsy
Whole body energy metabolism while awake | 1 and 2 days after circadian misalignment and matched times in control arm
  Measured by indirect calorimetry
Sleeping metabolic rate | 1.5 days after circadian misalignment and matched time in control arm
  Measured by indirect calorimetry
Skeletal muscle mtDNA | 1 and 2 days after circadian misalignment and matched times in control arm
  Measured by qPCR
Skeletal muscle mRNA | 1 and 2 days after circadian misalignment and matched times in control arm
  Measured by qPCR and Western Blotting
Skeletal muscle proteins | 1 and 2 days after circadian misalignment and matched times in control arm
  Measured by Western Blotting
Metabolic compounds in the blood (e.g. glucose, insulin, FFA's, Triglycerides, cholesterol) | 1 and 2 days after circadian misalignment and matched times in control arm
Core-body-temperature | 1 day after circadian misalignment and matched time in control arm
  Measured by a telemetric pill
Peripheral skin temperature | 1 day after circadian misalignment and matched time in control arm
  Measured by skin temperature sensors
Central skin temperature | 1 day after circadian misalignment and matched time in control arm
  Measured by skin temperature sensors
Heart rate | 1 day after circadian misalignment and matched time in control arm
  Measured by heart rate monitor

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Schrauwen, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University, Maastricht, Netherlands